CLINICAL TRIAL: NCT05351346
Title: A Study Comparing the Efficacy and Safety of Genotype-guided R-CHOP-X Versus R-CHOP in Patients With Diffuse Large B-Cell Lymphoma
Brief Title: Genotype-guided Treatment in DLBCL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: West China Hospital, Sichuan (Unknown); Qilu Hospital of Shandong University (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Second Hospital of Anhui Medical University (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Soochow University (Other); China-Japan Friendship Hospital (Other); Tongji Hospital (Other); Beijing Hospital (Other Government); The Second Affiliated Hospital of Dalian Medical University (Other); Zhujiang Hospital (Other); The First Affiliated Hospital of Anhui Medical University North District (Unknown); Hunan Cancer Hospital (Other); Liaoning Cancer Hospital & Institute (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Cancer Hospital Affiliated to Xinjiang Medical University (Unknown); The First Affiliated Hospital of Xiamen University (Other); The First Affiliated Hospital of Nanchang University (Other); LanZhou University (Other); Central South University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Yunnan Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Fujian Medical University Union Hospital (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Gansu Cancer Hospital (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); RenJi Hospital (Other); Shandong Cancer Hospital and Institute (Other); Affiliated Cancer Hospital of Harbin Medical University (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); Fudan University (Other); Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Pekcing Union Medical College (Unknown); Affiliated Hospital of Nantong University (Other); Yunnan First People's Hospital (Unknown); Shanxi Province Cancer Hospital (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Beijing Tongren Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); Harbin Institute of Hematology (Unknown); The First Affiliated Hospital of Guangzhou Medical University (Other); Affiliated Hospital of Guilin Medical College (Unknown); Air Force Military Medical University, China (Other); Affiliated Zhongshan Hospital of Dalian University (Other); Yantai Yuhuangding Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUIDANCE-02
Record Dates: First submitted 2022-04-24; First posted 2022-04-28 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; orelabrutinib; Lenalidomide; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-CHOP-X (Experimental): Patients in R-CHOP-X group will receive rituximab 375 mg/m² IV on day 1, cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 2, and prednisone 100 mg/day PO on days 2-6 of every 21-day cycle for the first cycle. For the remaining 5 cycles, they will receive orelabrutinib 150 mg/day PO on days 1-21, or lenalidomide 25 mg/day PO on days 2-11, or decitabine 10 mg/m² IV on days -5 to -1 followed by standard R-CHOP of every 21-day cycle.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Orelabrutinib; Drug: Lenalidomide; Drug: Decitabine
- R-CHOP (Active Comparator): Patients in R-CHOP group will receive rituximab 375 mg/m² IV on day 1, cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² iv, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 2, and prednisone 100 mg/day PO on days 2-6 of every 21-day cycle for 6 cycles.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Rituximab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Cyclophosphamide — Cyclophosphamide IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Doxorubicin — Doxorubicin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Vincristine — Vincristine IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Prednisone — Prednisone PO will be administered as per the schedule specified in the respective arm.
Drug: Orelabrutinib — Orelabrutinib PO will be administered as per the schedule specified in the respective arm.
  Arms: R-CHOP-X
Drug: Lenalidomide — Lenalidomide PO will be administered as per the schedule specified in the respective arm.
  Arms: R-CHOP-X
Drug: Decitabine — Decitabine IV infusion will be administered as per the schedule specified in the respective arm.
  Arms: R-CHOP-X

SUMMARY:
A multicenter, prospective, randomized, open-label, controlled trial to evaluate the efficacy and safety of genotype-guided targeted agents plus rituximab-cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP-X) versus rituximab-cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in patients with diffuse large B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diffuse large B-cell lymphoma (without central nervous system involvement)
* Availability of archival or freshly collected tumor tissue before study enrolment
* International Prognostic Index (IPI) score of 2-5 or 1 with bulky disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Life expectancy greater than or equal to (>/=) 6 months
* The patient or his or her legal representative must provide written informed consent prior to any special examination or procedure for the research

Exclusion Criteria:

* Previous chemotherapy.
* Previous stem cell transplantation.
* History of malignancies except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrolled cardio- and cerebro-vascular disease, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
* Patients with central nervous system (CNS) lymphoma
* Primary mediastinal large B-cell lymphoma
* Left ventricular ejection fraction<50%
* Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

  1. Neutrophils<1.5×10^9/L
  2. Platelets<75×10^9/L (Platelets<50×10^9/L in case of bone marrow involvement)
  3. ALT or AST is 2 times higher than the upper limits of normal (ULN), AKP and bilirubin are 1.5 times higher than the ULN.
  4. Creatinine is 1.5 times higher than the ULN.
* HIV-infected patients
* Positive test results for chronic hepatitis B and hepatitis C infection
* Patients with psychiatric disorders or patients who are known or suspected to be unable to fully comply with the study protocol
* Pregnant or lactation
* Require treatment with strong/moderate CYP3A inhibitors or inducers.
* Inability to swallow capsules or presence of diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, post-bariatric surgery, inflammatory bowel disease and complete or incomplete intestinal obstruction
* Other medical conditions determined by the researchers that may affect the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Complete response rate | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 4 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No